CLINICAL TRIAL: NCT04164901
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-Controlled Study of AG-881 in Subjects With Residual or Recurrent Grade 2 Glioma With an IDH1 or IDH2 Mutation
Brief Title: Study of Vorasidenib (AG-881) in Participants With Residual or Recurrent Grade 2 Glioma With an IDH1 or IDH2 Mutation (INDIGO)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AG881-C-004; 2019-002481-13 (EudraCT Number); 2024-512961-15-00 (EU CTIS Number)
Record Dates: First submitted 2019-11-11; First posted 2019-11-15 (Actual); Results first posted 2023-11-24 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Grade 2 Glioma; Residual Glioma; Recurrent Glioma
Keywords: AG-881
MeSH Terms: conditions — Glioma | interventions — vorasidenib

STUDY DESIGN:
Intervention Model Description: Participants randomized in a 1:1 allocation (vorasidenib vs Placebo)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vorasidenib (Experimental): Vorasidenib 40 mg, continuous daily dosing.
  Interventions: Drug: Vorasidenib
- Matching Placebo (Placebo Comparator): Matching placebo 40 mg, continuous daily dosing.
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Vorasidenib — Vorasidenib oral film-coated tablets
  Other Names: AG-881
  Arms: Vorasidenib
Drug: Matching Placebo — Matching Placebo oral tablets
  Arms: Matching Placebo

SUMMARY:
Study AG881-C-004 is a phase 3, multicenter, randomized, double-blind, placebo-controlled study comparing the efficacy of vorasidenib to placebo in participants with residual or recurrent Grade 2 glioma with an IDH1 or IDH2 mutation who have undergone surgery as their only treatment. Participants will be required to have central confirmation of IDH mutation status prior to randomization. Approximately 340 participants are planned to be randomized 1:1 to receive orally administered vorasidenib 40 mg QD or placebo.

ELIGIBILITY:
Key Inclusion Criteria:

* Be at least 12 years of age and weigh at least 40 kg.
* Have Grade 2 oligodendroglioma or astrocytoma per WHO 2016 criteria.
* Have had at least 1 prior surgery for glioma (biopsy, sub-total resection, gross-total resection), with the most recent surgery having occurred at least 1 year (-1 month) and not more than 5 years (+3 months) before the date of randomization, and no other prior anticancer therapy, including chemotherapy and radiotherapy and not be in need of immediate chemotherapy or radiotherapy in the opinion of the Investigator.
* Have confirmed IDH1 (IDH1 R132H/C/G/S/L mutation variants tested) or IDH2 (IDH2 R172K/M/W/S/G mutation variants tested) gene mutation status disease by central laboratory testing during the Prescreening period and available 1p19q status by local testing (eg, fluorescence in situ hybridization [FISH], comparative genomic hybridization [CGH] array, sequencing) using an accredited laboratory.
* Have MRI-evaluable, measurable, non-enhancing disease, as confirmed by the BIRC.
* Have a Karnofsky Performance Scale (KPS) score (for participants ≥16 years of age) or Lansky Play Performance Scale (LPPS) score (for participants <16 years of age) of ≥80%.

Key Exclusion Criteria:

* Have had any prior anticancer therapy other than surgery (biopsy, sub-total resection, gross-total resection) for treatment of glioma including systemic chemotherapy, radiotherapy, vaccines, small-molecules, IDH inhibitors, investigational agents, laser ablation, etc.
* Have features assessed as high-risk by the Investigator, including brainstem involvement either as primary location or by tumor extension, clinically relevant functional or neurocognitive deficits due to the tumor in the opinion of the Investigator (deficits resulting from surgery are allowed), or uncontrolled seizures (defined as persistent seizures interfering with activities of daily life AND failed 3 lines of antiepileptic drug regimens including at least 1 combination regimen).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2020-01-05 (Actual); Primary Completion 2022-09-06 (Actual); Study Completion 2028-05 (Estimated)

CONTACTS AND LOCATIONS:
Locations (84):
- United States (40):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope, Duarte, California
  - University of California San Diego, La Jolla, California
  - UCLA Oncology Center, Los Angeles, California
  - University of California Irvine - Hospital, Orange, California
  - University of California San Francisco, San Francisco, California
  - Stanford Cancer Center, Stanford, California
  - University of Colorado Hospital - Anschutz Cancer Pavilion, Aurora, Colorado
  - Yale University, Yale Cancer Center, New Haven, Connecticut
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Sylvester Comprehensive Cancer Center - University of Miami Hospital and Clinics, Miami, Florida
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Maine Medical Partners Neurology, Scarborough, Maine
  - John Hopkins Cancer Center, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Metro Minnesota Community Oncology, Minneapolis, Minnesota
  - Mayo Comprehensive Cancer, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Tennessee Oncology, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - The University of Utah, Huntsman Cancer Hospital, Salt Lake City, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington
- Canada (5):
  - BC Cancer Agency, Vancouver, British Columbia
  - London Health Sciences Centre, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - McGill University Health Center, Montreal, Quebec
- France (4):
  - Centre Hospitalier Universitaire de Lille, Lille
  - Hôpital Pierre Wertheimer, Lyon
  - Hopitaux de La Timone, Marseille
  - Hospitalier Pitié Salpétrière, Paris
- Germany (4):
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Klinikum Mannheim Universitätsklinikum, Mannheim
- Israel (4):
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (5):
  - Azienda Ospedaliera Città della Salute e della Scienza di Torino, Turin, Piedmont
  - Ospedale Bellaria, Bologna
  - Istituto Oncologico Veneto - I.R.C.C.S., Padua
  - Istituto Nazionale Tumori Regina Elena, Roma
  - Istituto Clinico Humanitas, Rozzano
- Japan (9):
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Fujita Health University Hospital, Toyoake, Aichi-ken
  - Hiroshima University Hospital, Minami-Ku, Hiroshima
  - The University of Tokyo Hospital, Bunkyō-Ku, Tokyo
  - National Cancer Center Hospital, Chuo Ku, Tokyo
  - Kumamoto University Hospital, Kumamoto
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto
  - Kyoto University Hospital, Kyoto
  - Okayama University Hospital, Okayama
- Netherlands (3):
  - Haaglanden MC, Antoniushove, Leidschendam, South Holland
  - Erasmus Medical Center, Rotterdam
  - Universitair Medisch Centrum Utrecht, Utrecht
- Spain (3):
  - Hospital Universitario Vall d'Hebrón, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Switzerland (3):
  - Hôpitaux Universitaire de Genève, Geneva
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Universitätsspital Zürich, Zurich
- United Kingdom (4):
  - Freeman Hospital, Newcastle upon Tyne, England
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - Western General Hospital Edinburgh - PPDS, Edinburgh
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/

REFERENCES:
- [Result] Mellinghoff IK, van den Bent MJ, Blumenthal DT, Touat M, Peters KB, Clarke J, Mendez J, Yust-Katz S, Welsh L, Mason WP, Ducray F, Umemura Y, Nabors B, Holdhoff M, Hottinger AF, Arakawa Y, Sepulveda JM, Wick W, Soffietti R, Perry JR, Giglio P, de la Fuente M, Maher EA, Schoenfeld S, Zhao D, Pandya SS, Steelman L, Hassan I, Wen PY, Cloughesy TF; INDIGO Trial Investigators. Vorasidenib in IDH1- or IDH2-Mutant Low-Grade Glioma. N Engl J Med. 2023 Aug 17;389(7):589-601. doi: 10.1056/NEJMoa2304194. Epub 2023 Jun 4. PMID 37272516
- [Derived] Cloughesy TF, van den Bent MJ, Touat M, Blumenthal DT, Peters KB, Ellingson BM, Clarke JL, Mendez J, Yust-Katz S, Welsh L, Mason WP, Ducray F, Umemura Y, Nabors B, Holdhoff M, Hottinger AF, Arakawa Y, Sepulveda JM, Wick W, Soffietti R, Perry J, Giglio P, de la Fuente M, Maher E, Bottomley A, Tron AE, Yi D, Zhao D, Pandya SS, Steelman L, Hassan I, Wen PY, Mellinghoff IK; INDIGO trial investigators. Vorasidenib in IDH1-mutant or IDH2-mutant low-grade glioma (INDIGO): secondary and exploratory endpoints from a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2025 Dec;26(12):1665-1675. doi: 10.1016/S1470-2045(25)00472-3. Epub 2025 Oct 29. PMID 41175888
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vorasidenib | Matching Placebo
Started (The participant flow data is based on the Full Analysis Set (FAS) which includes all subjects randomized, classified according to the randomized treatment arm.) | 168 (One subject in the vorasidenib arm withdrew consent prior to treatment. They are counted in the total number started.) | 163
Completed (As the study is still ongoing, the number of participants "Completed" reflects the number of participants who were still on study at the time of data collection for the purposes of this results submission.) | 164 | 159
Not Completed | 4 | 4
Not completed — Withdrawal by Subject | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vorasidenib | Matching Placebo | Total
Number analyzed (Participants) | 168 | 163 | 331
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (10.51) | 39.8 (9.53) | 40.4 (10.04)
Age, Customized [Count of Participants; unit: Participants]
  Participant Age: 12 to less than 16 years old | 0 | 0 | 0
  Participant Age: 16 to less than 18 years old | 0 | 1 | 1
  Participant Age: 18 to less than 40 years old | 76 | 87 | 163
  Participant Age: 40 to less than 65 years old | 90 | 74 | 164
  Participant Age: 65 years or older | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 77 | 144
  Male | 101 | 86 | 187
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 9 | 18
  Not Hispanic or Latino | 122 | 135 | 257
  Unknown or Not Reported | 37 | 19 | 56
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 1 | 0 | 1
  Race: Asian | 5 | 8 | 13
  Race: Black or African American | 2 | 1 | 3
  Race: Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  Race: White | 125 | 132 | 257
  Race: Other | 2 | 1 | 3
  Race: Not reported | 33 | 21 | 54
Region of Enrollment [Number; unit: participants]
  Canada | 9 | 7 | 16
  Netherlands | 5 | 5 | 10
  United States | 77 | 100 | 177
  Italy | 4 | 6 | 10
  United Kingdom | 7 | 10 | 17
  Israel | 25 | 16 | 41
  France | 20 | 12 | 32
  Switzerland | 8 | 1 | 9
  Germany | 7 | 2 | 9
  Spain | 6 | 4 | 10
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] — Population: Data was not available
  kg/m^2
    number analyzed (Participants) | 166 | 162 | 328
    (all) | 26.81 (5.748) | 26.52 (5.887) | 26.66 (5.810)

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from date of randomization to date of first documented radiographic PD (as assessed by the blinded independent review committee (BIRC) per modified Response Assessment for Neuro-oncology for Low-Grade Gliomas or date of death due to any cause, whichever occurs earlier.
Time Frame: Up to approximately 30 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vorasidenib | Matching Placebo
Number analyzed (Participants) | 168 | 163
months | 27.7 [17.0 to NA] — Data was not estimable (median survival time exceeds the longest observed or censored survival time as of the data cut-off date) | 11.1 [11.0 to 13.7]
Statistical Analysis 1: Comparison: Vorasidenib vs Matching Placebo; Test type: Superiority; p < 0.0000001, Kaplan-Meier; Cox Proportional Hazard = 0.39, 95% CI 2-sided [0.27 to 0.56]

2. Secondary Outcome: Time to Next Intervention (TTNI)
Description: TTNI is defined as the time from randomization to the initiation of the first subsequent anticancer therapy (including vorasidenib, for subjects randomized to placebo who subsequently cross over) or death due to any cause.
Time Frame: Up to approximately 3 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Matching Placebo: Matching placebo 40 mg, continuous daily dosing. Matching Placebo: Matching Placebo oral tablets
Arm/Group | Vorasidenib | Matching Placebo
Number analyzed (Participants) | 168 | 163
months | NA [NA to NA] — Data was not estimable (median survival time exceeds the longest observed or censored survival time as of the data cut-off date) | 17.8 [15.0 to NA] — Data was not estimable (median survival time exceeds the longest observed or censored survival time as of the data cut-off date)

3. Secondary Outcome: Tumor Growth Rate (TGR)
Description: Calculated as the mean of the percentage change in tumor volume every 6 months
Time Frame: every 6 months, up to 2 years and 9 months
Measure: Mean (95% Confidence Interval); unit: percent change
Arm/Group | Vorasidenib | Matching Placebo
Number analyzed (Participants) | 168 | 163
percent change | -2.5 [-4.7 to -0.2] | 13.9 [11.1 to 16.8]

4. Secondary Outcome: Objective Response (OR) as Assessed by the Blinded Independent Review Committee (BIRC)
Description: OR is defined as a best overall response (BOR) of Complete Response, Partial Rresponse, or minor Response as assessed by the BIRC per the modified Response Assessment in Neuro-oncology for Low-grade Gliomas (RANO-LGG).
Time Frame: approximatively 30 months
Measure: Count of Participants; unit: Participants
Arm/Group | Vorasidenib | Matching Placebo
Number analyzed (Participants) | 168 | 163
Participants | 18 | 4
Statistical Analysis 1: Comparison: Vorasidenib vs Matching Placebo; Test type: Superiority; p = 0.003, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 4.88, 95% CI 2-sided [1.56 to 15.25] — Odds ratio was calculated with placebo as the control (denominator)

5. Secondary Outcome: Complete Response (CR) and Partial Response (PR) by BIRC
Description: CR and PR is defined as a BOR of CR or PR as assessed by BIRC per the modified RANO-LGG
Time Frame: Approximatively 30 months
Measure: Count of Participants; unit: Participants
Arm/Group | Vorasidenib | Matching Placebo
Number analyzed (Participants) | 168 | 163
Participants | 2 | 0

6. Secondary Outcome: Time to Response (TTR) by BIRC
Description: TTR is defined as the time from the date of randomization to the date of first documented CR, PR, or mR by BIRC per the modified RANO-LGG
Time Frame: Approximatively 30 months
Population: The number of participants with CR, PR or mR was 18 and 4, respectively in the vorasidenib and placebo groups. The median time duration of response is analysed only on participants with response.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Vorasidenib | Matching Placebo
Number analyzed (Participants) | 18 | 4
months | 11.0 [6.0 to 13.4] | 6.9 [4.1 to 9.7]

7. Secondary Outcome: Time to CR+PR by BIRC
Description: Time to CR+PR is defined as defined as the time from the date of randomization to the date of first documented CR or PR for subjects with CR or PR per the modified RANO-LGG (by BIRC)
Time Frame: Approximatively 30 months
Population: The number of participants with CR or PR was 2 and 0, respectively in the vorasidenib and placebo groups. The median time duration of response is analysed only on participants with response.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Vorasidenib | Matching Placebo
Number analyzed (Participants) | 2 | 0
months | 9.6 [5.6 to 13.6] |

8. Secondary Outcome: Duration of Response (DoR)
Description: DoR is defined as the time from the date of first documented CR, PR, or mR to the date of death due to any cause or date of first documented radiographic Prgressive Disease, whichever occurred earlier
Time Frame: Approximatively 30 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vorasidenib | Matching Placebo
Number analyzed (Participants) | 18 | 4
months | 16.6 [2.8 to 16.6] | NA [NA to NA] — The median and confidence interval were estimated from Kaplan- Meier method. They were not estimable as very few participants experienced the event.

9. Secondary Outcome: Duration of CR+PR
Description: Duration of CR+PR is defined as the time from the date of first documented CR or PR to the date of death due to any cause or first documented radiographic PD, whichever occurred earlier
Time Frame: Approximatively 30 months
Population: The number of participants with CR or PR was 2 and 0, respectively in the vorasidenib and placebo groups. In the placebo group, no participants experienced the event.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vorasidenib | Matching Placebo
Number analyzed (Participants) | 2 | 0
months | 13.8 [NA to NA] — The median and confidence interval were estimated from Kaplan- Meier method. The confidence limits were not estimable as very few participants experienced the event. |

10. Secondary Outcome: Overall Survival (OS)
Description: OS wad defined as the time from the date of randomization to the date of death due to any cause or data cutoff.
Time Frame: Approximatively 30 months
Population: This is based off of the participants in the Safety Set, which includes all subjects that received one least one dose of treatment. The months of survival represent the time between randomization and the data cutoff point, since during the study there were no deaths.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vorasidenib | Matching Placebo
Number analyzed (Participants) | 167 | 163
months | NA [NA to NA] — Not estimable since there were no deaths during the study | NA [NA to NA] — Not estimable since there were no deaths during the study

11. Secondary Outcome: Progression-Free Survival (PFS) by the Investigator
Description: PFS as assessed by the Investigator per the modified RANO-LGG
Time Frame: Approximatively 30 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vorasidenib | Matching Placebo
Number analyzed (Participants) | 168 | 163
months | NA [27.1 to NA] — Data was not estimable (median survival time exceeds the longest observed or censored survival time as of the data cut-off date) | 14.1 [11.2 to 18.5]
Statistical Analysis 1: Comparison: Vorasidenib vs Matching Placebo; Test type: Superiority; p = 0.00000024, Kaplan-Meier; Cox Proportional Hazard = 0.35, 95% CI 2-sided [0.23 to 0.54]

12. Secondary Outcome: Health-Related Quality of Life (FACT-Br)
Description: Health-Related Quality of Life (HRQoL) Functional Assessment of Cancer Therapy-Brain (FACT-Br) is a 50-item measure comprising the following subscales: Physical Well-Being, Functional Well-Being, Emotional Well-Being, and Social Well-Being subscales from the FACT-General (FACT-G), with the addition of a 23-item brain tumor-specific subscale. These subscales are summed to provide a total score. The total score is given at the end of treatment and total scores range from 0 to 200. Higher scores indicate a better HRQoL
Time Frame: Approximatively 30 months
Population: The low number of participants is related to the measure performed at the end of treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Vorasidenib | Matching Placebo
Number analyzed (Participants) | 21 | 47
units on a scale | 150.8 (29.5) | 151.8 (31.09)

ADVERSE EVENTS:
Time Frame: Approximately 30 months
Description: All AEs were recorded starting at the first dose through 28 days after the last dose. After the 28-day follow-up period, only SAEs that were considered related to IMP were reported. The data below reflects the subjects assigned to Vorasidenib or placebo, prior to the placebo group being eligible to cross over to receive Vorasidenib, an option after the study was unblinded. AEs are based on the participants in the Safety Analysis Set, who received at least 1 dose of the treatment or placebo.
Groups:
- Vorasidenib: Vorasidenib 40 mg, continuous daily dosing.
  Vorasidenib: Vorasidenib oral film-coated tablets
  One subject in the vorasidenib arm withdrew consent prior to treatment and did not receive the study drug; as a consequence the number of subjects in this group is 167
- Matching Placebo: Matching placebo 40 mg, continuous daily dosing.
  Matching Placebo: Matching Placebo oral tablets
  The data reflects the subjects assigned to placebo, prior to the placebo group being eligible to cross over to receive Vorasidenib, which was an option after the study was unblinded.
Arm/Group | Vorasidenib | Matching Placebo
All-Cause Mortality (participants affected / at risk) | 0/167 | 0/163
Serious Adverse Events (participants affected / at risk) | 11/167 | 8/163
Other Adverse Events (participants affected / at risk) | 158/167 | 152/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vorasidenib (N=167) | Matching Placebo (N=163)
Seizure (Nervous system disorders) | 5 | 3
Encephalopathy (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 1
Toxic encephalopathy (Nervous system disorders) | 0 | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Postprocedural infection (Infections and infestations) | 1 | 0
Alanine immunotransferase increased (Investigations) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 2
Myocardial ischemia (Cardiac disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Hematoma (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vorasidenib (N=167) | Matching Placebo (N=163)
Headache (Nervous system disorders) | 45 | 44
Dizziness (Nervous system disorders) | 25 | 26
Seizure (Nervous system disorders) | 18 | 16
Paraesthesia (Nervous system disorders) | 11 | 10
Diarrhoea (Gastrointestinal disorders) | 41 | 27
Nausea (Gastrointestinal disorders) | 36 | 37
Constipation (Gastrointestinal disorders) | 21 | 20
Abdominal Pain (Gastrointestinal disorders) | 14 | 14
Vomiting (Gastrointestinal disorders) | 11 | 16
Alanine aminotransferase increased (Investigations) | 64 | 24
Aspartate aminotransferase increased (Investigations) | 48 | 13
Gamma-glutamyltransferase increased (Investigations) | 26 | 8
COVID-19 (Infections and infestations) | 55 | 47
Fatigue (General disorders) | 54 | 52
Asthenia (General disorders) | 9 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 | 15
Myalgia (Musculoskeletal and connective tissue disorders) | 12 | 10
Back Pain (Musculoskeletal and connective tissue disorders) | 10 | 9
Hyperglycaemia (Metabolism and nutrition disorders) | 16 | 7
Decreased appetite (Metabolism and nutrition disorders) | 15 | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 13 | 8
Insomnia (Psychiatric disorders) | 16 | 13
Anxiety (Psychiatric disorders) | 9 | 15
Depression (Psychiatric disorders) | 6 | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 7 | 9
Vision Blurred (Eye disorders) | 4 | 9
Hypertension (Vascular disorders) | 9 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-07-20): https://cdn.clinicaltrials.gov/large-docs/01/NCT04164901/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-04): https://cdn.clinicaltrials.gov/large-docs/01/NCT04164901/SAP_001.pdf